CLINICAL TRIAL: NCT00690391
Title: Analysis of Palliative Surgery in View of Quality of Life and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: PD Dr. Christoph Wullstein, PD Dr. Christoph Wullstein
Other Study IDs: PS2008
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-05

CONDITIONS: Cancer; Quality of Life
Keywords: surgery; prognostic; palliation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical observation: patients with cancer in a palliative setting and in need of surgical interventions

SUMMARY:
The purpose of this study is to define if palliative surgery in patients with cancer improves quality of life and prognosis.

DETAILED DESCRIPTION:
The purpose of this study is to find out if palliative surgery in patients with cancer improves quality of life and prognosis. There will be a scheduled assessment of quality of life and assessment of postoperative complications. prognostic scoring will be performed before surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of inoperable cancer
* planned surgery
* able to give interview
* written informed consent

Exclusion Criteria:

* unconsciousness
* psychiatric disorder
* not able to communicate in German

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with plannes surgery and cancer in he University hospital Frankfurt
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-05 (Estimated); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Wullstein, PD DR., Principal Investigator — Goethe University
Locations (1):
- University hospital Frankfurt, Frankfurt, Germany